CLINICAL TRIAL: NCT03864341
Title: ED-Home: A Pilot Feasibility Study of a Homelessness Prevention Intervention for Substance Using Emergency Department Patients
Brief Title: ED-Home Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-02040; K23DA039179 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: Housing Problems; Drug Use; Alcohol; Use, Problem
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homelessness Prevention Services (Experimental)
  Interventions: Behavioral: Referral to homelessness prevention services; Behavioral: Substance use services; Behavioral: Follow-up

INTERVENTIONS:
Behavioral: Referral to homelessness prevention services — Referral to Homebase homelessness prevention services offered by community-based organizations in NYC
Behavioral: Substance use services — Referral to substance use services (SBIRT and peer counselor/social work contact) available at Bellevue Hospital
Behavioral: Follow-up — Follow-up to assist participants in receiving homelessness prevention services

SUMMARY:
This is a single-arm pilot study to test the feasibility of homelessness prevention and substance use interventions to be delivered to at-risk patients in the Bellevue Hospital emergency department (ED). ED patients (n=40) found eligible for the study will complete a baseline assessment and receive referrals to appropriate services, with a final six-month follow-up assessment.

DETAILED DESCRIPTION:
ED patients found eligible for the study will complete a baseline survey and receive one-time, in person services at the time of the baseline/enrollment ED visit including referrals to homelessness prevention and substance use services, with a final six-month follow-up survey. Interim contacts at 7-10 days, 3 months, and 5 months will be used to assure intervention components were received and to confirm participant contact information.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient in the Bellevue Hospital Center ED.
* Be ≥18 years old.
* Screen positive for homelessness risk using a homelessness risk screening tool (HRST).
* Screen positive for unhealthy alcohol or drug use.
* Able to provide consent.

Exclusion Criteria:

* Medically (e.g., critically ill) or psychiatrically unstable.
* Unable to provide informed consent for other reason (e.g., cognitive deficit, profound intoxication).
* Incarcerated or in police custody.
* Unable to understand and speak English.
* Lives outside NYC and/or cannot give a NYC ZIP code.
* Already homeless (residing in a shelter or on the streets).
* Does not have a telephone where can be reached for follow-up.
* Has already received specialized peer navigator/addiction social worker services during current ED visit.
* Has already participated in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Doran, MD, MHS, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Homelessness Prevention Services
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Homelessness Prevention Services
Number analyzed (Participants) | 39
Age, Continuous [Mean (Full Range); unit: years] | 44 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 6
  More than one race | 1
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Potential Participants Approached Who Were Eligible for the Study
Time Frame: Month 6
Population: This feasibility endpoint is related to the percentage of potential participants approached who were eligible to participate in the study -- since the number of eligible people is greater than those who were enrolled, the total number of "participants" analyzed is greater than what is listed in the participant flow.
Measure: Number; unit: Percentage of Participants
Arm/Group | Homelessness Prevention Services
Number analyzed (Participants) | 2183
Percentage of Participants | 2.34

2. Primary Outcome: Percentage of Eligible Participants Who Agreed to Participate in the Study
Time Frame: Month 6
Population: This feasibility endpoint is related to the percentage of eligible people who agreed to participate in the study -- since the number of eligible people is greater than those who were enrolled, the total number of "participants" analyzed is greater than what is listed in the participant flow.
Measure: Number; unit: Percentage of Participants
Arm/Group | Homelessness Prevention Services
Number analyzed (Participants) | 51
Percentage of Participants | 78.43

3. Primary Outcome: Number of Participants Who Received Referrals for Homelessness Prevention and/or Substance Use Services
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Homelessness Prevention Services
Number analyzed (Participants) | 39
Participants | 39

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Homelessness Prevention Services
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03864341/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03864341/ICF_000.pdf